CLINICAL TRIAL: NCT00687960
Title: Effect of Resistant Starch Type 4 on Glycemia and Insulin Sensitivity in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: MGP Ingredients, Inc. (Industry)
Responsible Party: Mark Haub Ph.D., Department of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: KSU-HML-RSt2
Record Dates: First submitted 2008-05-22; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Hyperglycemia
Keywords: Diabetes; Diet; Fiber; Age
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Resistant Starch Type 4-Raw
  Interventions: Dietary Supplement: Resistant starch type 4 - raw
- 2 (Experimental): Resistant Starch Type 4-cooked
  Interventions: Dietary Supplement: Resistant Starch Type 4 - Cooked
- 3 (Active Comparator): Puffed wheat
  Interventions: Dietary Supplement: Puffed Wheat
- 4 (Placebo Comparator): Dextrose
  Interventions: Dietary Supplement: Dextrose

INTERVENTIONS:
Dietary Supplement: Resistant starch type 4 - raw — Dose: 80g bar containing Resistant Starch Type 4 - raw
  Arms: 1
Dietary Supplement: Resistant Starch Type 4 - Cooked — Dose: 80g bar containing Resistant Starch Type 4 - cooked
  Arms: 2
Dietary Supplement: Dextrose — Dose: 7 oz of oral glucose tolerance beverage
  Arms: 4
Dietary Supplement: Puffed Wheat — Dose: 80g bar containing puffed wheat cereal
  Arms: 3

SUMMARY:
This study tested the effects of resistant starch type 4 on blood sugar and hunger in young adults with Type 2 diabetes.

DETAILED DESCRIPTION:
To measure the blood glucose response, after an overnight fast, blood samples were collected before eating and at 15, 30, 45, 60, 90, and 120 minutes after each each bar. The incremental area under the curve was used to calculate the glycemic index and insulin sensitivity via minimal model.

ELIGIBILITY:
Inclusion Criteria:

* Apparently Healthy (not diagnosed with disease)
* Young Adults (18-35)

Exclusion Criteria:

* Diagnosed with diabetes or other metabolic disorders
* Allergies to Wheat
* Non-smokers

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Post-Prandial Metabolism | Early morning

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haub, Ph.D., Principal Investigator — Department of Human Nutrition
Locations (1):
- Kansas State University, Manhattan, Kansas, United States